CLINICAL TRIAL: NCT07047547
Title: A Prospective, Observational, Single-arm Study to Evaluate the Efficacy and Safety of Vericiguat in Patients With Chronic Kidney Disease and Heart Failure.
Brief Title: A Study of Real-world Events of Vericiguat in Patients With Chronic Kidney Disease and Heart Failure
Acronym: ESVGR-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, ShuangXin Liu, Chief Physician, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250624
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis Complication; Heart Failure
Keywords: Vericiguat; Heart failure; Hemodialysis Complication
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vericiguat (Experimental): Under the premise of ensuring safety, treat with a stable dose of Vericiguat 2.5mg PO QD for 2 weeks. After 2 weeks, increase the dose to 5mg PO QD. If blood pressure elevation occurs during the operation phase, the researchers suggest titrating or starting additional antihypertensive drugs, with a follow-up of 12 months. If the patient has tolerability issues (symptomatic hypotension or SBP<90 mmHg), the dose should be reduced or discontinued.
  Interventions: Drug: Vericiguat

INTERVENTIONS:
Drug: Vericiguat — Under the premise of ensuring safety, treat with a stable dose of Vericiguat 2.5mg PO QD for 2 weeks. After 2 weeks, increase the dose to 5mg PO QD. If blood pressure elevation occurs during the operation phase, the researchers suggest titrating or starting additional antihypertensive drugs, with a follow-up of 12 months. If the patient has tolerability issues (symptomatic hypotension or SBP<90 mmHg), the dose should be reduced or discontinued.

SUMMARY:
Chronic Kidney Disease often requires dialysis and other treatments to sustain life, and patients frequently suffer from heart failure, which exacerbates the disease burden. Research has shown that the incidence of heart failure is high among patients on dialysis, and the prognosis is poor. In recent years, there has been significant progress in the treatment of heart failure. Vericiguat, a novel sGC stimulator, can improve cardiac function and exercise tolerance, reduce the risk of cardiovascular death and hospitalization for heart failure, and has good tolerance. It has been included in relevant guidelines as a recommended drug. It has good tolerance in patients with renal insufficiency, and its therapeutic effect is consistent in patients with different levels of eGFR. However, there is a lack of prospective, randomized controlled studies targeting the special population of patients on dialysis. This study is a prospective, observational, single-arm study, planning to recruit 118 patients from June 2025 to June 2026. It aims to assess the efficacy and safety of Vericiguat in patients with heart failure on hemodialysis, to provide new evidence-based medical evidence for the treatment of heart failure in this special population, optimize the treatment strategy, and improve the prognosis and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The patient is aged between 18 and 80 years
* Suffering from chronic kidney disease (eGFR<90ml/min/1.73m², by CKD-EPI formula).
* They have chronic heart failure (NYHA class ≥II), with reduced ejection fraction, defined as LVEF≤50%.
* Their serum potassium level has been ≤4.8 mmol/L in the past month.
* For women of childbearing potential, the pregnancy test result is negative at the screening visit and they agree.
* Adequate contraceptive measures are taken.
* The patient's dialysis adequacy assessment has reached Kt/V >1.2, or URR>70%.
* The study protocol is implemented after being approved by the hospital ethics committee, and all patients voluntarily participate in this study

Exclusion Criteria:

* Acute renal failure.
* Systolic blood pressure below 90 mmHg at screening (systolic blood pressure less than 95 mmHg during interdialytic period).
* Isolated right heart failure due to pulmonary disease; the primary cause of dyspnea is due to non-cardiac, non-heart failure reasons, such as acute or chronic respiratory diseases.
* History of myocardial infarction or cerebrovascular event within the past 3 months.
* History of angioedema.
* Hemodialysis patients with dialysis frequency less than 3 times per week.
* Significant laboratory abnormalities at screening that interfere with the assessment of the safety or efficacy of the study drug (e.g., serum potassium > 5.5 mmol/L or < 3.5 mmol/L, serum sodium < 130 mmol/L, or alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of the normal range).
* History of kidney transplantation or planned kidney transplantation within the next 12 months.
* Use of medications for pulmonary arterial hypertension, such as sildenafil, during the study period.
* Known allergy to the study treatment (active substance or excipients).
* Any other disease or treatment that makes the patient ineligible to participate in this study or to complete the entire planned study period (e.g., active malignancy or other diseases that limit life expectancy to less than 12 months).
* Pregnant or breastfeeding during the study period, or intending to become pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction(LVEF) | 12weeks
  Change from baseline in left ventricular ejection fraction(LVEF)between baseline and end of study
Left ventricular ejection fraction (LVEF) | 12weeks
  Change from baseline in left ventricular ejection fraction (LVEF) between baseline and end of study

SECONDARY OUTCOMES:
N terminal proB type natriuretic peptide (NT-prpBNP) | 12 weeks
  Blood samples will be collected for analysis of concentration of N terminal pro B type natriuretic pel proBNP) every 2 weeks
Left ventricular end diastolic volume (LVEDV) | 12 weeks
  LVEDV is measured as baseline and after 12 weeks follow-up.
Left atrial volume (LAV) | 12 weeks
  LAVis measured as baseline and after 12 weeks follow-up.
The ratio of mitral early diastolic blood flow peak and mitral annulus velocity (E/E') | 12 weeks
  E/E' is measured as baseline and after 12 weeks follow-up.
Pulmonary Artery Pressure | 12 weeks
  Pulmonary Artery Pressure is measured as baseline and after 12 weeks follow-up.
Concentration of high-sensitivity serum troponin T | 12 weeks
  Blood samples will be collected for analysis of concentration of serum troponin every 4 weeks.
Minnesota Heart Failure Quality of Life Questionnaire (LiHFe) | 12 weeks
  Change in health status is assessed using the disease-specific Minnesota Heart Failure Quality of L Questionnaire.
Systolic and diastolic blood pressure | 12 weeks
  Systolic and diastolic blood pressure will be measured every 2 weeks.
Electrocardiogram(ECG) | 12 weeks
  ECG QT Interval analysis was performed at baseline and 12 weeks follow-up.
Estimated glomerular filtration rate(eGFR) | 12 weeks
  changes in estimated glomerular filtration rate(eGFR)

OTHER OUTCOMES:
Neprilysin | 12 weeks
  The concentration of Neprilysis is measured by Human Neprilysin ELISA Kit as baseline and after 12 weeks following up

CONTACTS AND LOCATIONS:
Overall Officials: Shuangxin Liu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China